CLINICAL TRIAL: NCT02948972
Title: Impact of Complete Surgery of Colorectal Deep Infiltrating Endometriosis on Fertility: Complete Surgery + IVF Versus IVF (ENDOFERT)
Brief Title: Impact of Complete Surgery of Colorectal Deep Infiltrating Endometriosis on Fertility
Acronym: ENDOFERT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015_02; 2015 A01536-43 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-10-04; First posted 2016-10-31 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Endometriosis; Infertility
Keywords: deep infiltrating endometriosis; endometriosis surgery; In vitro fertilization
MeSH Terms: conditions — Endometriosis; Infertility | interventions — Fertilization in Vitro; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- complete surgery (Experimental): Prior surgery 3 months before IVF followup 1, 6 12 and 24 month after surgery
  Interventions: Procedure: complete surgery; Procedure: In vitro fertilization without surgery
- In vitro fertilization without surgery (Active Comparator): IVF without endometriosis surgery follow up 6, 12 and 24 month after inclusion.
  Interventions: Procedure: In vitro fertilization without surgery

INTERVENTIONS:
Procedure: complete surgery — complete surgery of colorectal deep infiltrating endometriosis
  Arms: complete surgery
Procedure: In vitro fertilization without surgery — IVF without endometriosis surgery

SUMMARY:
The ENDOFERT Study is an open, multicenter, randomized, parallel-group, controlled trial. This study includes patients presenting colorectal DIE and infertility. Patients will be randomized in two parallel-groups; one group underwent complete surgery of colorectal DIE prior to ART and the other group underwent ART alone (ratio 1:1)

ELIGIBILITY:
Inclusion Criteria:

* Primary and secondary infertility
* Indication for IVF
* Persistent pain related to endometriosis with analgesic medical treatment failure
* Persistent pain including at least one of the following digestive symptoms related to endometriosis: Dyschesia / Sub-occlusive syndrome / Rectal bleeding / Painful defecation
* Colorectal deep infiltrating endometriosis : Whatever lesion size / With at least rectal serosal involvement / Confirmed by MRI and 1 different investigation: vaginal ultrasound echography or coloscopic CT scan or rectal endoscope ultrasound
* Eligible for DIE surgery

Exclusion Criteria:

* Contraindication to pregnancy or to IVF
* Viral risk
* Previous IVF cycle(s)
* Previous colorectal surgery
* Need of myomectomy during surgery
* The use of oocytes donor

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-11-17 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy after 2 IVF cycles | At the end of the 2nd IVF cycle (therefore at 6 weeks after each embryo transfer)
  Clinical pregnancy is defined as pregnancy at 6 weeks of gestation with ultrasound echographic confirmation.
  An IVF cycle is defined as the transfer of all the embryos created via IVF after 1 oocytes puncture until a pregnancy confirmation or until the failure of the last embryo transfer. 2 embryos are transferred for each transfer steps.
  The length of one cycle depend on the number of embryo transfer steps. It is usually between 2 and 9 months.

SECONDARY OUTCOMES:
predictive factors | At the end of the 2nd IVF cycle
  The expected predictive factors observed according to the fecundity status after 2 IVF cycles
  An IVF cycle is defined as the transfer of all the embryos created via IVF after 1 oocytes puncture until a pregnancy confirmation or until the failure of the last embryo transfer. 2 embryos are transferred for each transfer steps.
  The length of one cycle depend on the number of embryo transfer steps. It is usually between 2 and 9 months.
Clinical pregnancy rate after 1st IVF cycle | At the end of the 1st IVF cycle (therefore at 6 weeks after each embryo transfer)
  Clinical pregnancy is defined as pregnancy at 6 weeks of gestation with ultrasound echographic confirmation.
  An IVF cycle is defined as the transfer of all the embryos created via IVF after 1 oocytes puncture until a pregnancy confirmation or until the failure of the last embryo transfer. 2 embryos are transferred for each transfer steps.
  The length of one cycle depend on the number of embryo transfer steps. It is usually between 2 and 9 months.
Clinical pregnancy rate per embryo transferred | At the end of the 2nd IVF cycle (therefore at 6 weeks after each embryo transfer)
  Clinical pregnancy is defined as pregnancy at 6 weeks of gestation with ultrasound echographic confirmation.
  An IVF cycle is defined as the transfer of all the embryos created via IVF after 1 oocytes puncture until a pregnancy confirmation or until the failure of the last embryo transfer. 2 embryos are transferred for each transfer steps.
  The length of one cycle depend on the number of embryo transfer steps. It is usually between 2 and 9 months.
The IVF complication | 24 months after surgery or inclusion in "IVF without surgery" group
  rate of hyperstimulation, superinfection, worsening of pain and hospitalization related to IVF procedures in each group.
perioperative complications | 24 months after surgery
  Complications rate of perioperative surgical excision according to the CLAVIEN-DINDO grading system and to the Comprehensive Complication Index
The cumulative IVF cycle cancellation rate | At the end of the 2nd IVF cycle
  The cumulative IVF cycle cancellation rate in each group.
  An IVF cycle is defined as the transfer of all the embryos created via IVF after 1 oocytes puncture until a pregnancy confirmation or until the failure of the last embryo transfer. 2 embryos are transferred for each transfer steps.
  The length of one cycle depend on the number of embryo transfer steps. It is usually between 2 and 9 months.
Endometriosis Health Profile -5 (short form / EHP5) | during inclusion, 6, 12 and 24 months after surgery or inclusion in "IVF without surgery" group
  Evolution of quality life scores in each group
Gastrointestinal Quality of Life Index. (GIQLI) | during inclusion, 6, 12 and 24 months after surgery or inclusion in "IVF without surgery" group
  Evolution of quality life scores in each group
Short Form (36) Health Survey _ SF 36 | during inclusion, 6, 12 and 24 months after surgery or inclusion in "IVF without surgery" group
  Evolution of quality life scores in each group
Evaluation of hemorrhagic, digestive, urinary symptoms Dysmenorrhea and pains not related to menstruation | during inclusion, 6, 12 and 24 months after surgery or inclusion in "IVF without surgery" group
  * Dysmenorrhea and pains not related to menstruation will be evaluated by Visual Analog Scale (VAS)
  * Evolution of the hemorrhagic, digestive and urinary symptoms at 6, 12 and 24 months
Knowles Eccersley Scott Symptom (KESS) score | during inclusion, 6, 12 and 24 months after surgery or inclusion in "IVF without surgery" group
  Evolution of the bowel function score KESS

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Collinet, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (5):
- France (5):
  - CHU, Clermont-Ferrand
  - Hôpital Jeanne de Flandres, CHRU, Lille
  - AP-HP, Hôpital Tenon, Paris
  - CHU, Poissy
  - CHU, Rouen

IPD SHARING:
Plan to Share IPD: No